CLINICAL TRIAL: NCT03058133
Title: Neural Correlates of Multimodal Face/Voice Processing in a Gender Task.
Brief Title: Gender in Face-Voice Integration
Acronym: Face-Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0674
Record Dates: First submitted 2017-02-08; First posted 2017-02-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: fMRI, perception, face-voice processing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fMRI study (Other)
  Interventions: Other: fMRI study

INTERVENTIONS:
Other: fMRI study — Functional brain activations of face-voice processing during a gender task

SUMMARY:
Bayesian models of perception represent a promising approach to describe information processing by the brain. Predictive coding hypothesizes a process in which top-down expectations are continuously compared across multiple hierarchical levels with bottom-up sensory inputs and the differences or error signals are propagated in a bottom-up direction. The investigators hypothesize that strong expectations, are best investigated in expert processes such as face and voice recognition in humans. Individuals in complex social systems need to extract socially relevant information in a fast and efficient manner; hence, the majority of humans constitute face, voice and gender experts. Nevertheless, linking such combined abilities to brain activity with regards to the predictive coding hypothesis has not been attempted.Our results suggest asymmetric contributions of visual and auditory signals to the gender classification task. This sensitive psychophysical procedure is implemented in a decoding approach using fMRI and multi-voxel pattern analysis (MVPA). The investigators plan to test whether cortical areas implicated in processing auditory and visual gender signals show similar asymmetries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, right-handed
* No neurological antecedent
* Signed informed consent

Exclusion Criteria:

* Pregnant women
* Volunteers with MRI contraindications: persons using a pacemaker or insulin pump, persons with a metallic prosthesis or an intracerebral clip, as well as claustrophobic subjects, neurosensory stimulator or implantable defibrillator, cochlear implants, body Foreign ferromagnetic ocular or cerebral close to nerve structures, agitation of the subject (non-cooperating or agitated subjects), ventriculoperitoneal neurosurgical bypass valves, dental apparatus.
* Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights or liberty, as well as persons of legal age protected by law.
* Participants refusing to be informed of the results of the medical examination (inclusion).
* Participants refusing to be informed of the possible detection of an anomaly.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Identify neural correlates (fMRI) of face / voice interaction in a gender classification task | Maximum 90 days between inclusion of the subject and the 1st fMRI session (1h1 / 2). Then maximum 90 days before the 2nd session (1h1 / 2).
  Classical functional analyses (GLM) and advanced statistical analyses of brain activations (BrainVoyager and Matlab softwares).
Identify neural correlates (fMRI) of face / voice respective contribution in a gender classification task | Maximum 90 days between inclusion of the subject and the 1st fMRI session (1h1 / 2). Then maximum 90 days before the 2nd session (1h1 / 2).
  Classical functional analyses (GLM) and advanced statistical analyses of brain activations

CONTACTS AND LOCATIONS:
Overall Officials: Alain NICOLAS, MD, Principal Investigator — Le VINATIER
Locations (1):
- Le VINATIER, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbatecola C, Kennedy H, Knoblauch K. Directed attention influences optimality of top-down and bottom-up multi-modal perceptual integration. Sci Rep. 2025 Jul 16;15(1):25742. doi: 10.1038/s41598-025-09542-6. PMID 40670460
- [Background] Abbatecola C, Gerardin P, Beneyton K, Kennedy H, Knoblauch K. The Role of Unimodal Feedback Pathways in Gender Perception During Activation of Voice and Face Areas. Front Syst Neurosci. 2021 May 28;15:669256. doi: 10.3389/fnsys.2021.669256. eCollection 2021. PMID 34122023
- [Background] Gerardin P, Kourtzi Z, Mamassian P. Prior knowledge of illumination for 3D perception in the human brain. Proc Natl Acad Sci U S A. 2010 Sep 14;107(37):16309-14. doi: 10.1073/pnas.1006285107. Epub 2010 Aug 30. PMID 20805488
- [Background] Wacongne C, Changeux JP, Dehaene S. A neuronal model of predictive coding accounting for the mismatch negativity. J Neurosci. 2012 Mar 14;32(11):3665-78. doi: 10.1523/JNEUROSCI.5003-11.2012. PMID 22423089
- [Background] Pegado F, Comerlato E, Ventura F, Jobert A, Nakamura K, Buiatti M, Ventura P, Dehaene-Lambertz G, Kolinsky R, Morais J, Braga LW, Cohen L, Dehaene S. Timing the impact of literacy on visual processing. Proc Natl Acad Sci U S A. 2014 Dec 9;111(49):E5233-42. doi: 10.1073/pnas.1417347111. Epub 2014 Nov 24. PMID 25422460
- [Background] Markov NT, Ercsey-Ravasz M, Van Essen DC, Knoblauch K, Toroczkai Z, Kennedy H. Cortical high-density counterstream architectures. Science. 2013 Nov 1;342(6158):1238406. doi: 10.1126/science.1238406. PMID 24179228
- [Background] Charrier C, Knoblauch K, Maloney LT, Bovik AC, Moorthy AK. Optimizing multiscale SSIM for compression via MLDS. IEEE Trans Image Process. 2012 Dec;21(12):4682-94. doi: 10.1109/TIP.2012.2210723. Epub 2012 Jul 30. PMID 22868568
- [Background] Gerardin P, Devinck F, Dojat M, Knoblauch K. Contributions of contour frequency, amplitude, and luminance to the watercolor effect estimated by conjoint measurement. J Vis. 2014 Apr 10;14(4):9. doi: 10.1167/14.4.9. PMID 24722563